CLINICAL TRIAL: NCT05740293
Title: Post-approval Study of New Enrolment Patients Undergoing Bilateral Treatment With the VisuMax SMILE Procedure
Status: Completed | Type: Observational
Sponsor: Carl Zeiss Meditec, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: VisuMax-2018-PAS01
Record Dates: First submitted 2023-02-07; First posted 2023-02-23 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Myopia; Astigmatism
MeSH Terms: conditions — Myopia; Astigmatism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Procedure: VisuMax SMILE procedure for the reduction or elimination of myopia with astigmatism — Bilateral treatment with the approved VisuMax SMILE procedure for the reduction or elimination of myopia with astigmatism.

SUMMARY:
The objective of the post-approval study (PAS) is to assess patient experience of visual symptoms 6 months after bilateral treatment with the VisuMax SMILE procedure as measured by a patient questionnaire.

DETAILED DESCRIPTION:
This is a prospective, multicenter, single arm, open-label, observational study of newly enrolled patients undergoing bilateral treatment with the approved SMILE procedure for the reduction or elimination of myopia with astigmatism. Patients complete a self-administered patient questionnaire preoperatively and 6 months postoperatively. Each patient's preoperative status is serving as the control for postoperative endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for the approved VisuMax SMILE procedure according to the Professional Use Information, i.e.
* Spherical refractive error (in minus cylinder format) from -1.00 D through -10.00 D;
* Refraction spherical equivalent not greater in magnitude than 10.00 D;
* Minimum age of 22 years;
* Documentation of stable manifest refraction over the past year as demonstrated by a change in sphere and cylinder of ≤ 0.50 D in magnitude.
* Good candidate for SMILE based on the surgeon's assessment of medical and ophthalmic health, cognitive function, and physical and social limitations
* Intended bilateral SMILE treatment for the correction of myopia with astigmatism (-0.75 to -3.00 D)
* Both eyes targeted for the full distance manifest spherocylindrical refraction
* Fluent English in speaking and reading
* Willingness and ability to return for 6-month postoperative examination
* Signed informed consent

Exclusion Criteria:

* Presence of any of the contraindications of the approved SMILE procedure for the reduction or elimination of myopia with astigmatism, i.e.
* a residual stromal bed thickness that is less than 250 microns from the corneal endothelium;
* abnormal corneal topographic findings, e.g. keratoconus, pellucid marginal degeneration;
* ophthalmoscopic signs of progressive or unstable myopia or keratoconus (or keratoconus suspect);
* irregular or unstable (distorted/not clear) corneal mires on central keratometry images;
* severe dry eye;
* active eye infection or inflammation;
* recent herpes eye infection or problems resulting from past infection;
* active autoimmune disease or connective tissue disease;
* uncontrolled diabetes;
* uncontrolled glaucoma.
* Previous treatment with any form of refractive surgery

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will enroll and treat a maximum of 171 patients undergoing bilateral treatment with the approved SMILE procedure for the reduction or elimination of myopia with astigmatism from six (6) to ten (10) investigational sites in the U.S.A.
Sampling Method: Non-Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-08-25 (Actual)

PRIMARY OUTCOMES:
Development of clinically relevant visual symptoms via questionnaire responses | 6 months
  * Proportion of subjects that developed "very" or "extremely" bothersome visual symptoms from preoperative (with optical correction) to 6 months postoperatively (without optical correction)
  * Proportion of subjects that developed difficulty performing daily activities (2 highest categories) due to visual symptoms from preoperative (with optical correction) to 6 months postoperatively (without optical correction)

SECONDARY OUTCOMES:
Resolution of clinically relevant visual symptoms via questionnaire responses | 6 months
  * Proportion of subjects that showed resolution of "very" or "extremely" bothersome visual symptoms from preoperative (with optical correction) to 6 months postoperatively (without optical correction)
  * Proportion of subjects that showed resolution of difficulty performing daily activities (2 highest categories) due to visual symptoms from preoperative (with optical correction) to 6 months postoperatively (without optical correction)
Development and resolution of all visual symptoms via questionnaire responses | 6 months
  * Proportion of subjects that developed visual symptoms from preoperative (with optical correction) to 6 months postoperatively (without optical correction)
  * Proportion of subjects that showed resolution of visual symptoms from preoperative (with optical correction) to 6 months postoperatively (without optical correction)
Dry eye via questionnaire responses | 6 months
  * Proportion of subjects that developed dry eye symptoms as compared to their preoperative status (OSDI score from normal at preoperative to abnormal at 6 months; categorized according to Miller et al. 2010)
  * Proportion of subjects that showed resolution of dry eye symptoms as compared to their preoperative status (OSDI score from abnormal at preoperative to normal at 6 months; categorized according to Miller et al. 2010)
Satisfaction via questionnaire responses | 6 months
  * Proportion of patients satisfied with their vision after the SMILE procedure (who responded "completely satisfied", "very satisfied", or "somewhat satisfied" to the corresponding questionnaire item)
  * Proportion of patients satisfied with the SMILE procedure (based on a score ≥ 40 in the corresponding 8-item questionnaire domain)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Vold Vision, Fayetteville, Arkansas
  - IQ Laser Vision, Rowland Heights, California
  - Discover Vision Centers, Leawood, Kansas
  - Goel Vision, Columbia, Maryland
  - Cleveland Eye Clinic, Brecksville, Ohio
  - Parkhurst NuVision, San Antonio, Texas
  - Northwest Eye Surgeons, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No